CLINICAL TRIAL: NCT05593094
Title: A Phase 1 Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics (PK), and Efficacy of ZN-A-1041 Enteric Capsules as a Single Agent or in Combination in Patients With HER2-Positive Advanced Solid Tumors
Brief Title: A Phase 1 Trial of ZN-A-1041 Enteric Capsules or Combination in Participants With Human Epidermal Growth Factor Receptor 2 (HER2)-Positive Advanced Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: XO45189; ZN-A-1041-101-US (Other: Suzhou Zanrong Pharma Limited); 2023-508459-37-00 (EU CTIS Number)
Record Dates: First submitted 2022-10-17; First posted 2022-10-25 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Advanced Solid Tumors; HER2-positive Breast Cancer
Keywords: Phase 1; Advanced Solid Tumors; HER2 postive; Brain metastases; Herceptin; Perjeta; PHESGO; First Line; 1st Line
MeSH Terms: conditions — Brain Neoplasms | interventions — Ado-Trastuzumab Emtansine; Trastuzumab; pertuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- 1a: ZN-A-1041 (Experimental): Phase 1a:
  Participants will receive escalating doses of ZN-A-1041 orally twice a day (BID) at pre-defined dosing regimens to determine the maximum tolerated dose (MTD).
  Interventions: Drug: ZN-A-1041
- 1b: ZN-A-1041 + T-DM1 3.6 mg/kg iv. (Experimental): Phase 1b Arm1:
  1. If the maximum tolerated dose (MTD) of ZN-A-1041 is identified in Phase 1a study: The 2 tentative dose levels of ZN-A-1041 are MTD-1 (Level 1) and MTD (Level 2).
  2. If the MTD is still not reached at the maximum dose level in Phase 1a study, the maximum dose level of ZN-A-1041 in Phase 1a will be used in Phase 1b study.
  Interventions: Drug: ZN-A-1041 + T-DM1 3.6 mg/kg iv. for Phase 1b
- 1b: ZN-A-1041 + T-Dxd 5.4 mg/kg iv. (Experimental): Phase 1b Arm2:
  1. If the MTD of ZN-A-1041 is identified in Phase 1a study: The 2 tentative dose levels of ZN-A-1041 are MTD-1 (Level 1) and MTD (Level 2).
  2. If the MTD is still not reached at the maximum dose level in Phase 1a study, the maximum dose level of ZN-A-1041 in Phase 1a will be used in Phase 1b study.
  Interventions: Drug: ZN-A-1041 + T-Dxd 5.4 mg/kg iv. for Phase 1b
- 1b: ZN-A-1041 + PHESGO / Herceptin plus Perjeta (Experimental): Phase 1b Arm3:
  1. If the MTD of ZN-A-1041 is identified in Phase 1a study: The 2 tentative dose levels of ZN-A-1041 are MTD-1 (Level 1) and MTD (Level 2).
  2. If the MTD is still not reached at the maximum dose level in Phase 1a study, the maximum dose level of ZN-A-1041 in Phase 1a will be used in Phase 1b study.
  Interventions: Drug: ZN-A-1041 + PHESGO / Herceptin plus Perjeta injection for Phase 1b
- 1c: ZN-A-1041 + T-DM1 3.6 mg/kg iv. (Experimental): Phase 1c Arm1:
  The recommended dose combination for Phase 1c will be determined by the Investigator and the Sponsor based on the data from Phase 1b.
  Interventions: Drug: ZN-A-1041 + T-DM1 3.6 mg/kg iv. for Phase 1c
- 1c: ZN-A-1041 + T-Dxd 5.4 mg/kg iv. (Experimental): Phase 1c Arm2:
  The recommended dose combination for Phase 1c will be determined by the Investigator and the Sponsor based on the data from Phase 1b.
  Interventions: Drug: ZN-A-1041 + T-Dxd 5.4 mg/kg iv. for Phase 1c
- 1c: ZN-A-1041 + Herceptin plus Perjeta/PHESGO (Experimental): Phase 1c Arm3:
  The recommended dose combination for Phase 1c will be determined by the Investigator and the Sponsor based on the data from Phase 1b.
  Interventions: Drug: ZN-A-1041 + PHESGO / Herceptin plus Perjeta injection for Phase 1c

INTERVENTIONS:
Drug: ZN-A-1041 — ZN-A-1041: escalating doses orally BID at pre-defined dosing regimens to determine the MTD
  Other Names: ZN-A-1041 Enteric Capsules
  Arms: 1a: ZN-A-1041
Drug: ZN-A-1041 + T-DM1 3.6 mg/kg iv. for Phase 1b — ZN-A-1041: BID via oral administration T-DM1: 3.6 mg/kg given as an intravenous infusion on the first day of each treatment cycle, once every 3 weeks (21-day cycle)
  Other Names: ZN-A-1041 Enteric Capsules
  Arms: 1b: ZN-A-1041 + T-DM1 3.6 mg/kg iv.
Drug: ZN-A-1041 + T-Dxd 5.4 mg/kg iv. for Phase 1b — ZN-A-1041: BID via oral administration T-DXd: 5.4 mg/kg given as an intravenous infusion on the first day of each treatment cycle, once every 3 weeks (21-day cycle)
  Other Names: ZN-A-1041 Enteric Capsules
  Arms: 1b: ZN-A-1041 + T-Dxd 5.4 mg/kg iv.
Drug: ZN-A-1041 + PHESGO / Herceptin plus Perjeta injection for Phase 1b — ZN-A-1041: BID via oral administration PHESGO dose is 600 mg pertuzumab/600 mg trastuzumab/2000 unites hyaluronidase every 3 weeks for subcutaneous administrations (21-day cycle) Perjeta is 420 mg administered as an intravenous infusion Herceptin is 6 mg/kg administered as an intravenous infusion
  Other Names: ZN-A-1041 Enteric Capsules
  Arms: 1b: ZN-A-1041 + PHESGO / Herceptin plus Perjeta
Drug: ZN-A-1041 + T-DM1 3.6 mg/kg iv. for Phase 1c — ZN-A-1041: BID via oral administration T-DM1: intravenous infusion on the first day of each treatment cycle, once every 3 weeks (21-day cycle)
  Other Names: ZN-A-1041 Enteric Capsules
  Arms: 1c: ZN-A-1041 + T-DM1 3.6 mg/kg iv.
Drug: ZN-A-1041 + T-Dxd 5.4 mg/kg iv. for Phase 1c — ZN-A-1041: BID via oral administration T-DXd: intravenous infusion on the first day of each treatment cycle, once every 3 weeks (21-day cycle)
  Other Names: ZN-A-1041 Enteric Capsules
  Arms: 1c: ZN-A-1041 + T-Dxd 5.4 mg/kg iv.
Drug: ZN-A-1041 + PHESGO / Herceptin plus Perjeta injection for Phase 1c — ZN-A-1041: BID via oral administration PHESGO: every 3 weeks for subcutaneous administrations (21-day cycle) Perjeta: intravenous infusion Herceptin: intravenous infusion
  Other Names: ZN-A-1041 Enteric Capsules
  Arms: 1c: ZN-A-1041 + Herceptin plus Perjeta/PHESGO

SUMMARY:
This will be a Phase 1, multicenter, open-label trial to evaluate the safety, tolerability, PK and efficacy of ZN-A-1041 as a monotherapy or in combination in participants with HER2-positive advanced solid tumors with or without brain metastases.

The study will consist of three phases: Phase 1a (dose escalation with ZN-A-1041 monotherapy), Phase 1b (dose escalation with ZN-A-1041 combination therapy) and Phase 1c (dose expansion with ZN-A-1041 combination therapy).

DETAILED DESCRIPTION:
This study is composed of three parts designed to evaluate the safety and efficacy of ZN-A-1041 in participants with HER2-positive advanced solid tumors.

Phase 1a (Monotherapy Dose Escalation): In this first phase, participants will receive ZN-A-1041 alone. The study will begin with a low dose of ZN-A-1041, which will be gradually increased in new groups of participants to find the highest dose that can be given safely. This will establish the recommended dose for further study.

Phase 1b (Combination Dose Escalation): In the second phase, the study will evaluate the safety of giving ZN-A-1041 together with established standard-of-care therapies for HER2-positive breast cancer. Participants will be enrolled into one of three combination arms to receive ZN-A-1041 with either T-DM1, T-DXd, or a pertuzumab/trastuzumab-based regimen. This phase will identify the recommended dose for these combination therapies.

Phase 1c (Combination Dose Expansion): In the final phase, additional participants will be enrolled to receive ZN-A-1041 at the recommended combination doses identified in Phase 1b. This will allow for a more thorough evaluation of the safety and preliminary efficacy of these treatment regimens.

Throughout the study, participants will undergo screening, treatment, and follow-up periods to collect comprehensive data on the safety, tolerability, pharmacokinetics, and anti-tumor activity of ZN-A-1041, both as a single agent and in combination.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Life expectancy of at least 6 months, as determined by the investigator
* Histologically or cytologically confirmed with unresectable or metastatic HER2-positive advanced solid tumors
* Must be relapsed or refractory after prior treatment for metastatic disease that included a taxane and trastuzumab or must have received first-line induction therapy for advanced disease a pertuzumab plus trastuzumab-based regimen or a T-DXd-based regimen
* Participants with new, untreated, progressive, or stable brain metastases are eligible

Exclusion Criteria:

* Participation in any other clinical study involving an investigational drug or device within 4 weeks prior to the first dose of study treatment
* Any intracranial lesion (brain metastasis) that requires immediate local therapy, such as surgery or radiation, or systemic corticosteroids at the time of enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2020-09-03 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
The Incidence of Treatment-emergent Adverse Events of ZN-A-1041 as a Monotherapy in Phase 1a | 23 days
  Dose at which no more than one out of six participant at the same dose level experiences a probable drug-related DLT.
The Incidence of Treatment-emergent Adverse Events of ZN-A-1041 in Combination with T-DM1 or with T-DXd, or in Combination with PHESGO or Herceptin plus Perjeta | 21 days
  Dose at which no more than one out of six participant at the same dose level experiences a probable drug-related DLT.
RP2D | Through study completion, an average of 1 year
  To evaluate the safety of ZN-A-1041 in combination with T-DM1 or with T-DXd, or in combination with PHESGO or Herceptin plus Perjeta in participants on the RP2D.

SECONDARY OUTCOMES:
Plasma, Urine and Potentially Cerebrospinal Fluid (CSF) Level of ZN-A-1041 and its Main Metabolites | From baseline to cycle 9 (each cycel is 21 days)
  To assess the PK of ZN-A-1041 and its major metabolites.
Serum Level of Combination Drugs in Phase 1c | Through study completion, an average of 2 year
  To assess the serum concentration of combination drugs.
Anti-drug Antibodies (ADAs) Evaluation in Phase 1c | Through study completion, an average of 2 year
  To assess the incidence of ADAs.
Overall Response Rate (ORR) | Through study completion, an average of 2 year
  The preliminary efficacy of ZN-A-1041 as a monotherapy or combination in Phase 1a, Phase 1b and 1c.
Progression Free Survival (PFS) | Through study completion, an average of 2 year
  The preliminary efficacy of ZN-A-1041 as a monotherapy or combination in Phase 1a, Phase 1b and 1c.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (36):
- United States (8):
  - Arizona Clinical Research Center, Inc.;Hematology Oncology Physicians - Aoa, Tucson, Arizona
  - TOI Clinical Research, Cerritos, California
  - UCSF Helen Diller Family CCC, San Francisco, California
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan Hospital, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Duke University School of Medicine, Durham, North Carolina
  - MD Anderson Cancer Center, Houston, Texas
- Australia (2):
  - Geelong Hospital, Geelong, Victoria
  - Sunshine Hospital, St Albans, Victoria
- France (7):
  - EDOG - Institut Claudius Regaud - PPDS, Toulouse, Haute-Garonne
  - Centre Georges Francois Leclerc, Dijon
  - Centre Oscar Lambret, Lille
  - Centre Léon Bérard Centre Régional de Lutte Contre Le Cancer Rhône Alpes, Lyon
  - Institut Paoli-Calmettes, Marseille
  - Institut de Cancerologie de l Ouest, Saint-Herblain
  - Gustave Roussy, Villejuif
- Italy (3):
  - Istituto Romagnolo per lo Studio dei Tumori Dino Amadori - IRST S.r.l - PPDS, Parma, Emilia-Romagna
  - Asst Papa Giovanni XXIII, Bergamo, Lombardy
  - Fondazione Policlinico Universitario A Gemelli-Rome, Magnago, Lombardy
- Auckland City Hospital, Auckland, New Zealand
- Spain (13):
  - Instituto de Investigacion Oncologica Vall dHebron (VHIO) - EPON, Argentona, Barcelona
  - Hospital Clinico Universitario de Santiago, Santiago de Compostela, LA Coruna
  - Hospital Universitario Ramon y Cajal, A Gudiña, Orense
  - Hospital Universitario Virgen del Rocio, Las Cabezas de San Juan, Sevilla
  - Instituto Oncologico Dr. Rosell-Hospital Universitari Dexeus-Grupo Quironsalud, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitario de Jaen, Jaén
  - Hospital Beata Maria Ana, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Virgen Macarena, Seville
  - Fundacion Instituto Valenciano de Oncologia (IVO), Valencia
  - Hospital Clinico Universitario de Valencia, Valencia
- United Kingdom (2):
  - The Christie, Manchester, Lancashire
  - Clatterbridge Cancer Centre, Liverpool, Merseyside

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing